CLINICAL TRIAL: NCT03273179
Title: Cerebral Venous Sinus Thrombosis: Re-exploration of Clinical Assessment
Brief Title: Cerebral Venous Sinus Thrombosis: Re-exploration of Clinical Assessment Scales
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming, Professor, Capital Medical University
Other Study IDs: CVST-RCAS
Record Dates: First submitted 2017-09-03; First posted 2017-09-06 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Cerebral Venous Sinus Thrombosis; CSF Pressure Increased; Papilledema
Keywords: cerebral venous sinus thrombosis; CSF pressure; modified Rankin Scale; papilledema; NIHSS
MeSH Terms: conditions — Intracranial Hypertension; Papilledema

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a single-center, retrospective, open-label study. This study is planned to investigate the accuracy of mRS and NIHSS, comparing with the accuracy of CSF pressure and papilledema grade in assessing cerebral venous sinus thrombosis.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of CVST by head MRI, DSA or MRV onset of CVST within one month

Exclusion Criteria:

* unable to complete examinations unable to complete follow-ups

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All individual with confirmed diagnosis of CVST are eligible for this research
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-04-01 (Estimated); Study Completion 2018-07-01 (Estimated)

PRIMARY OUTCOMES:
baseline CSF pressure | baseline
  CSF pressure at baseline
baseline mRS | baseline
  mRS at baseline
baseline papilledema grade | baseline
  Frisen grade of papilledema at baseline

SECONDARY OUTCOMES:
baseline NIHSS | baseline
  NIH Stroke Scale at baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital Capital Medical University, Beijing, China